CLINICAL TRIAL: NCT02335307
Title: Implementing Genomics in Practice (IGNITE) Proof of Concept Study: Genotyping in Family Medicine Clinics
Acronym: IGNITE
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400501 - N; U01HG007269-02 (NIH); OCR14741 (Other: Universiy of Florida)
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: Pain; CYP2D6
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — genotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients will continue to receive their current pain management therapy. In addition, a pain assessment questionnaire will be administered at baseline and 3 months.
  Interventions: Other: Pain assessment questionnaire
- Implementation: Patients will undergo CYP2D6 genotyping, with results entered into the medical record to assist the physician with prescribing pain medication. In addition, a pain assessment questionnaire will be administered at baseline and 3 months.
  Interventions: Genetic: CYP2D6 genotyping; Other: Pain assessment questionnaire
- Physician assessment: At the end of the study, a 20-item survey will be administered to physicians who treated patients enrolled in the study. The survey will assess whether having CYP2D6 genotype results is useful to inform prescribing decisions for pain medication from the physician's perspective.
  Interventions: Other: Physician assessment

INTERVENTIONS:
Genetic: CYP2D6 genotyping — CYP2D6 genotype results and an interpretive report will be placed in the electronic medical record to assist the physician with prescribing medication for pain management.
  Groups: Implementation
Other: Pain assessment questionnaire — A pain assessment questionnaire will be administered at baseline and 3 months.
  Other Names: PROMIS questionnaire
  Groups: Control; Implementation
Other: Physician assessment — 20-item survey administered to physicians treating patients enrolled in the study
  Groups: Physician assessment

SUMMARY:
This study will examine the effect of having genotype information on pain management and pain control for patients treated in family medicine clinics. This study will also examine physician-perceived usefulness of genotype information. Patients will be enrolled from family medicine clinics serving as either implementation sites or control sites. Patients from implementation sites will undergo genotyping, while those from control sites will not by genotyped.

DETAILED DESCRIPTION:
Codeine and tramadol are opioid analgesics that depend on cytochrome P450 2D6 (CYP2D6) for bioactivation to morphine and O-desmethyltramadol, respectively. Morphine and O-desmethyltramadol have much greater affinity for the opioid receptor and thus are more powerful analgesics.

Individuals with genotypes associated with low CYP2D6 activity (poor metabolizers) are unable to convert sufficient amounts of codeine or tramadol to their active metabolites and may fail to derive sufficient pain relief. At the opposite extreme, individuals with genotypes associated with increased CYP2D6 activity (ultra-rapid metabolizers) are at risk for serious toxicity with usual codeine or tramadol doses.

The CYP2D6 genotype also has implications for response to other drugs, such as tricyclic antidepressants (TCAs), which are commonly used for neuropathic pain.

Patients will be recruited from family medicine clinics, serving as either implementation sites or control sites. Patients from implementation sites will undergo CYP2D6 genotyping, with results placed in the medical record to assist with prescribing of pain medications. Pain medications prescribed from baseline to 3 months will be assessed through medical record review. A pain assessment questionnaire will be administered to patients enrolled from both sites at baseline and 3 months.

At the end of the study, a 20-item survey will be administered to physicians at the implementation sites. We will assess whether having CYP2D6 genotype results is useful to inform prescribing decisions for pain medication from the physician's perspective.

We will also assess medicines prescribed to patients enrolled from both sites over the 12-month period after enrollment from medical record review and determine the number of patients who were prescribed a medication that has genetic information in its FDA-approved label.

ELIGIBILITY:
Inclusion Criteria:

* Treated in family medicine clinic
* History of pain for at least 3 months
* Prescribed medication for pain relief

Exclusion Criteria:

* Pain for less than 3 months
* Not currently prescribed any medication for pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from family medicine clinics serving as either implementation sites or control sites for pain mangement.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Change in overall pain score (Patient Reported Outcomes Measurement Information System (PROMIS) | Change from baseline to 3 months
  Patient Reported Outcomes Measurement Information System (PROMIS) measures will be used to assess pain intensity, physical functioning, and emotional functioning. There are 10 subscales on the PROMIS questionnaire that address the domains of pain, pain functioning, and emotional functioning. At least 4 (and up to 30) items are used to derive a score for each subscale. A computer adaptive version of the questionnaire based on item response theory will be used to administer the survey. A score of 0 to 100 based on survey responses will be resulted for each subscale.

SECONDARY OUTCOMES:
Change in pain medication | Change from baseline to 3 months
  Change in pain medication will be evaluated in several manners: change in the opiate prescribed, change from an opiate to a non-opiate; and change in dose of the opiate prescribed
Change in pain score of pain intensity (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | Change from baseline to 3 months
  Patient Reported Outcomes Measurement Information System (PROMIS) subscale for pain intensity, with the score ranging from 0 to 100 resulting.
Change in pain score of physical functioning (Patient Reported Outcomes Measurement Information System (PROMIS) subscale) | Change from baseline to 3 months
  Patient Reported Outcomes Measurement Information System (PROMIS) subscales for physical functioning include pain function, pain interference, pain behavior, sleep disturbance, and sleep-related impairment. A score of 0 to 100 based on survey responses will be resulted for each subscale.
Change in pain score of emotional functioning | Change from baseline to 3 months
  Patient Reported Outcomes Measurement Information System (PROMIS) subscales for emotional functioning include fatigue, anxiety, depression, and anger. A score of 0 to 100 based on survey responses will be resulted for each subscale.
Physician perceived usefulness of genetic information (survey) | 3 months
  Survey will be administered to physicians with patients in the study to assess the effect of having genotype information on their prescribing decisions.
Medications prescribed with pharmacogenetic implications (Percent of patients with at least one other drug (besides an opioid) where genotype information might be useful for prescribing) | 12 months
  Percent of patients with at least one other drug (besides an opioid) where genotype information might be useful for prescribing

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Cavallari, PharmD, Principal Investigator — University of Florida
Locations (11):
- United States (11):
  - Archer Family Health Care, Archer, Florida
  - UF Health Spring Hill Pain Management, Gainesville, Florida
  - UF Health Family Medicine: Hampton Oaks, Gainesville, Florida
  - UF Health Internal Medicine - Tower Hill, Gainesville, Florida
  - UF Health Family Medicine: Haile Plantation, Gainesville, Florida
  - UF Health Family Medicine: Main Street, Gainesville, Florida
  - UF Health Internal Medicine-Medical Plaza, Gainesville, Florida
  - UF Health Family Medicine: Eastside, Gainesville, Florida
  - UF Health Family Medicine - Old Town, Old Town, Florida
  - Oviedo Family Health Center, Oviedo, Florida
  - ProHealth Family Physicians, Saint Cloud, Florida

IPD SHARING:
Plan to Share IPD: Yes
The consent form has an addendum for NIH dbGaP. Participants who agree will have their deidentified results shared to dbGaP. Those who do not agree will not have their results shared.

REFERENCES:
- [Background] Crews KR, Gaedigk A, Dunnenberger HM, Leeder JS, Klein TE, Caudle KE, Haidar CE, Shen DD, Callaghan JT, Sadhasivam S, Prows CA, Kharasch ED, Skaar TC; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium guidelines for cytochrome P450 2D6 genotype and codeine therapy: 2014 update. Clin Pharmacol Ther. 2014 Apr;95(4):376-82. doi: 10.1038/clpt.2013.254. Epub 2014 Jan 23. PMID 24458010